CLINICAL TRIAL: NCT04566926
Title: A 3-Part, Randomized, Placebo-controlled, Double-blind, Single Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-64140284 in Healthy Male Participants
Brief Title: A Study of JNJ-64140284 in Healthy Male Participants
Acronym: AMPAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108866; 2020-002616-40 (EudraCT Number); 64140284EDI1005 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2020-09-24; First posted 2020-09-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: Cohort 1 (Placebo or JNJ-64140284) (Experimental): Participants will receive matching placebo in Treatment A or JNJ-64140284 (as formulation 1) in Treatment B or JNJ-64140284 (as formulation 2) in Treatment C on Day 1 under fasted condition. Participants will receive treatment in either of the 6 treatment sequences (ABC, BCA, CAB, CBA, ACB or BAC) in Period 1, 2, or 3 under fasted condition. Each period is separated by washout period of 5 days.
  Interventions: Drug: JNJ-64140284; Drug: Placebo
- Part 1: Cohort 2 (Placebo or JNJ-64140284) (Experimental): Participants will receive matching placebo (Treatment D) or JNJ- 64140284 (as formulation 1) in Treatment E or JNJ-64140284 (as formulation 2) in Treatment F. Participants will receive treatment in either of 6 treatment sequence (DEF, EFD, FDE, FED, DFE or EDF) in Period 1, 2, or 3 under fed condition. Each period is separated by washout period of 5 days.
  Interventions: Drug: JNJ-64140284; Drug: Placebo
- Part 2: Cohorts 1-7 (JNJ-64140284 or Placebo) (Experimental): Participants will receive JNJ 64140284 formulation 1 or 2 or matching placebo under fasting condition in Cohorts 1 to 7 on Day 1.
  Interventions: Drug: JNJ-64140284; Drug: Placebo
- Part 3: Cohorts 1-2 (JNJ-64140284 or placebo) (Experimental): Participants will receive JNJ-64140284 formulation 1 or 2 or matching placebo under fed condition in Cohorts 1 to 2 on Day 1.
  Interventions: Drug: JNJ-64140284; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64140284 — Participant will receive JNJ-64140284 formulation 1 or 2 under fasting or fed condition.
Drug: Placebo — Participant will receive matching placebo.

SUMMARY:
The purpose of the study is to investigate and compare the pharmacokinetic (PK) profiles of a single dose of two solid dosage formulations of JNJ-64140284 in plasma and urine in healthy male participants under fed and fasting conditions; and to investigate the safety and tolerability of two solid dosage formulations of JNJ 64140284 versus placebo after single oral dose administration in healthy male participants under fed and fasting conditions in Part 1; to investigate the safety and tolerability of JNJ-64140284 versus placebo after single oral dose administration (or 1 divided dose, if applicable) (ascending dose levels) in healthy male participants; and to characterize the PK of a single dose (or 1 divided dose, if applicable) of JNJ-64140284 in plasma in healthy male participants in Part 2; and to investigate the effect of food on the PK of a single (or 1 divided dose, if applicable) therapeutic relevant dose of JNJ 64140284 in healthy male participants; and to investigate the safety and tolerability of JNJ-64140284 versus placebo after single oral dose administration at a therapeutic relevant dose (or 1 divided dose, if applicable) in fed conditions in Part 3.

ELIGIBILITY:
Inclusion criteria:

* Participant has a body mass index (BMI) between 18.0 and 29.9 kilograms per square meters (kg/m^2) inclusive
* Participant must be healthy on the basis of clinical laboratory tests. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed. The participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must be healthy on the basis of physical and neurological examination, medical history, vital signs, and 12-lead Electrocardiogram (ECG) (means of triplicate ECG, incl. QTcF less than or equal to [<=] 450 milliseconds [msec] for males). Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable
* A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person and must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 3 months after receiving the last dose of study intervention
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion criteria:

* Participant has history of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Participant has a Left Bundle Branch Block (LBBB), atrioventricular (AV) Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator (ICD)
* Participant has a history of suicidal ideation or a family history of suicide
* Participant has a history of major depressive disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti HCV at screening

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Part 1: Plasma Concentration of JNJ-64140284 | Pre-dose, Day 1, 2, 3 and Day 4
  Plasma samples will be analyzed to determine concentrations of JNJ-64140284 under fed and fasting conditions using a validated, specific and sensitive liquid chromatography-mass spectrometry (LC-MS/MS).
Part 1: Urine Concentration of JNJ-64140284 | Pre-dose, Day 1, 2, 3 and Day 4
  Urine samples will be analyzed to determine concentrations of JNJ-64140284 in renal clearance.
Part 2: Plasma Concentration After Single Dose Administration of JNJ-64140284 | Pre-dose, Day 1, 2, 3 and Day 4
  Plasma samples will be analyzed to determine concentrations of JNJ-64140284 under fed and fasting conditions using a validated, specific and sensitive liquid chromatography-mass spectrometry (LC-MS/MS).
Part 3: Ratio of Area Under Plasma Concentration Curve (AUC) and Maximum Plasma Concentration (Cmax) | Pre-dose, Day 1, 2, 3 and Day 4
  Ratio of geometric means for pharmacokinetics (PK) parameters (AUCs and Cmax) of JNJ 64140284 (fed versus fasted condition) will be analyzed to determine the food effect.
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability: Part 1, Part 2, and Part 3 | Up to 1.5 years
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An adverse event does not necessarily have a causal relationship with the intervention. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.

SECONDARY OUTCOMES:
Bond & Lader Visual Analogue Scale (VAS) Score: Part 1 and Part 2 | Day -1, 1, 2 and Day 3
  The VAS is a participant rated scale, made up of 16 (items) pairs of alternative descriptors of mood and attention at either end of a 10-centimeter (cm) line. The item score ranges from 0 to 100, with a high score reflecting a high level of anxiety, sedation or dysphoria.
Karolinska Sleepiness Scale (KSS) Score: Part 1 and Part 2 | Day -1, 1, 2 and Day 3
  The KSS is a participant-reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep' (9).
Body Sway | Day -1, 1, 2 and Day 3
  Body sway will be used to measure body movements, providing a measure of postural stability. The method has been used to demonstrate effects of sleep deprivation, alcohol, and benzodiazepines. It will be measured either using a stabilometric platform or a pot string meter based on the Wright ataxiameter.
Part 2: Pharmacodynamics (PD) as Assessed by Cognitive Test Battery: Detection Task (DET) | Day -1, 1, 2 and Day 3
  DET is a measure of psychomotor function. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: Identification Task (IDN) | Day -1, 1, 2 and Day 3
  IDN is a measure of attention. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: One Card Learning Task (OCL) | Day -1, 1, 2 and Day 3
  OCL is a measure of visual learning. The test measures accuracy of performance; arcsine transformation of the square root of the proportion of correct responses. Higher score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: One Back Task (ONB) | Day -1, 1, 2 and Day 3
  ONB is a measure of working memory. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: Groton Maze Learning Test (GMLT) | Day -1, 1, 2 and Day 3
  GMLT is a measure of executive function and spatial learning. The test measures total number of errors made while locating and learning 28 step pathway hidden beneath a 10*10 grid on 5 consecutive trials during a single session. Lower score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: International Shopping List Test (ISLT) | Day -1, 1, 2 and Day 3
  The ISLT is a measure of verbal learning. The test measures total number of correct responses remembering the word list on 3 consecutive trials at a single assessment. Higher score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: International Shopping List Test delayed (ISLT-D) | Day -1, 1, 2 and Day 3
  ISLT-D is a measure of delayed verbal memory. The test measures total number of correct responses recalling the word list learned initially. Higher score indicates better performance.
Part 2: PD as Assessed by Cognitive Test Battery: Groton Maze Learning Test delayed (GMLT-D) | Day -1, 1, 2 and Day 3
  GMLT delayed recall is a measure of delayed spatial memory. The test measures number of errors made while locating 28 step pathway hidden beneath a 10*10 grid after a delay. Lower score indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (1):
- SGS Life Science Services, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency